CLINICAL TRIAL: NCT05689307
Title: Validation Study With a Non-CE Marked Medical Device (MD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siva Health AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIVA-VS2
Record Dates: First submitted 2023-01-06; First posted 2023-01-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SIVA-MVP (Experimental): Wearable cough detection device with a corresponding smartphone application and charging device.
  Interventions: Device: SIVA-MVP

INTERVENTIONS:
Device: SIVA-MVP — Participants receive a small, wearable data recorder, wear it during the day and charge it on the nightstand during sleep for 14x24 hours. The encrypted, recorded segments are uploaded to a server. The server provides a secure environment where the segments are decrypted after receiving the required keys from the patient's SIVA smartphone application. The decrypted segments are then classified as cough by a machine learning algorithm. Participants respond to questions on a smartphone once a day for additional context data. The audio data from the first 24 hours after the patient started wearing the device are used for the validation of the performance of the cough detection algorithm.

SUMMARY:
This interventional study aims to validate the cough detection device by automatically and continuously measuring the cough frequency with SIVA-MVP among chronic cough patients and in a real-world environment.

DETAILED DESCRIPTION:
After chronic cough diagnosis, the Principal Investigator (or his designee) will identify potentially eligible patients to participate in this study based on the predefined inclusion criteria.

The study will recruit patients with a cough that has lasted for at least 12 months and persistent for the previous 8 weeks with a diagnosis or suspicion of refractory chronic cough, or patients with a diagnosed asthma. A total of 50 patients will be enrolled in the study.

Patients who decide to participate will be entered into the study after obtaining their informed consent. They will receive the SIVA-MVP wearable and the associated accessories. They will be asked to rate their current cough severity on a visual analog scale (Cough Severity VAS) and fill in a Leicester Cough Questionnaire (LCQ) to assess the impact of cough on their quality of life. Participants will receive a second Cough Severity VAS and LCQ to fill at the end of the study and a return envelope.

Participants will receive standard care and be asked to wear SIVA-MVP on their chest during the day and charge it on the bedside during sleep for 14 days. Every evening, they will be prompted by the SIVA-MVP smartphone application to indicate the timing of their main meals.

On day 15, the study nurse will conduct a pre-scheduled phone interview with each participant. The phone interview will include instructing the patient to fill in the final Cough Severity VAS and LCQ, asking the questions of the Participant User Feedback Questionnaire, and instructing the patient to send the questionnaire forms and the SIVA-MVP wearable and the accessories back to the trial site using the return envelope. The Participant User Feedback Questionnaire will include ratings of wearing comfort, usability, and likeliness to wear for an extended period of time.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Adult men and women at the date of signing the Informed Consent Form
* Patients with a diagnosis or suspicion of refractory chronic cough or patients with a diagnosed asthma
* Attending the treatment procedure as an outpatient
* Comfortable with using a smartphone and willing to use an external iPhone daily for the duration of the study.
* Adequate communication in US English (all study documentation and SIVA-MVP will be set to English language only).

Exclusion Criteria:

* Unable to make the decision to participate in a clinical study (e.g., seriously ill or unconscious subject, or subject with a mental or intellectual disability)
* Inability to follow the procedures of the study, e.g., due to physical or intellectual impairment precluding informed consent or protocol adherence, psychological disorders (excluding depression) or dementia
* Use of any other medical device equipment (e.g., portable oxygen concentrator, artificial cardiac pacemaker, implantable cardioverter-defibrillator)
* Pregnancy: Female participants in child-bearing age without a negative pregnancy test (urine test). Female participants who are neither surgically sterilized / hysterectomized nor post-menopausal for longer than 2 years are considered to be of childbearing potential.
* Known or suspected non-compliance, drug or alcohol abuse
* Participation in another clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Performance of the SIVA-MVP cough detection device | First 24 hours
  Validation of a SIVA-MVP performance of detecting individual cough events in a target population over a 24-hour validation phase (first 24 hours after baseline visit). Sensitivity, specificity, and positive and negative predictive values contribute to a description of cough monitor performance.

SECONDARY OUTCOMES:
Wearing comfort | 2 weeks
  Wearing Comfort will be determined through quantitative analysis of questions in the Participant User Feedback Questionnaire measured with 5-level Likert Scale (Disagree, Somewhat disagree, Neither agree nor disagree, Somewhat agree, Agree).
Number of potential adverse events, serious adverse events, device deficiency and serious device deficiency | 2 weeks
  Device safety measured as the number of potential adverse events, serious adverse events, device deficiency and serious device deficiency.
Comparison of objectively recorded (device) data and subjectively reported (patient) data measured with Leicester Cough Questionnaire and Cough Severity VAS | At Baseline and at the end of 2 weeks
  Correlation of patient reported outcomes measured with Leicester Cough Questionnaire and Cough Severity Visual Analog Scale (VAS) with recorded cough frequency during 14x24h.
Wearing time | 2 weeks
  Effective wearing times per day as recorded by the device.
Effective reply rate | 2 weeks
  Effective reply rate of patients to questions for context information asked to them via the smartphone application
Cough frequency patterns | 2 weeks
  Degree of similarity between cough patterns of different days within one patient and between patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Bellingham Asthma, Allergy & Immunology Clinic, Bellingham, Washington, United States

IPD SHARING:
Plan to Share IPD: No